CLINICAL TRIAL: NCT01663454
Title: Computer Based Working Memory Training in Children With Cerebral Palsy, a Pilot Study
Brief Title: Working Memory Training in Children With Cerebral Palsy, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bhø_2011/2271
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Cerebral Palsy; Working Memory Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cogmed Robomemo working memory training (Experimental): Participants will complete 25 sessions (5 weeks) of Cogmed Robomemo (Pearson assessment) working memory training
  Interventions: Behavioral: Cogmed Robomemo working memory training

INTERVENTIONS:
Behavioral: Cogmed Robomemo working memory training — The Cogmed Robomemo program is designed as a computer game in which an animated robot gives different tasks to be solved by the child. The tasks have various degrees of difficulty adapted continuously throughout the intervention period to the performance of the individual child. The program is standardized in that each child receives the same set of tasks during the training period. The child will perform the training sessions at home using their own computer for about 35-40 minutes each day.

SUMMARY:
The purpose of this pilot study is to assist the preparation of a larger multi-center study. The main aim is to determine the feasibility of conducting computerized working memory training in a group of children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Born at term with unilateral spastic CP
* Born preterm with bilateral spastic CP

Exclusion Criteria:

* Children with Gross Motor Function Classification Scale (GMFCS) level V
* Severe visual or hearing impairments
* Photosensitive epilepsy

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in training index | Changes in training index is measured during 5 weeks of working memory training
  The training index is based on the user's best results from selected exercises in the program. The Start Index is calculated with the results from days 2 and 3, and the Max Index is calculated with the results from the two best days during the training period. The Index Improvement is calculated by subtracting the Start Index from the Max Index.

SECONDARY OUTCOMES:
Neuropsychological testing | baseline and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Beneventi, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway